CLINICAL TRIAL: NCT00972959
Title: A Prospective, Multicenter, Non-comparative, Open-label, Phase II Study to Evaluate the Effects of the Combination of Bortezomib/Dexamethasone/Zoledronic Acid on Bone Mineral Density, Bone Metabolism, Radiographically-detected Osteolytic Bone Lesions, Skeletal-related Events and Bone Pain in Patients With Multiple Myeloma Who Have Relapsed After 1-3 Prior Lines of Therapy
Brief Title: Effect of Combination of Bortezomib/Dexamethasone/Zoledronic Acid on Bone Disease in Patients With Multiple Myeloma Relapsed After 1-3 Prior Lines of Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Meletios A. Dimopoulos, Director of the clinic, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138MMY 2051
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; 1-3 Prior Lines of Therapy; bortezomib (Velcade); zoledronic acid (Zometa); Dexamethasone; bone mineral density; bone pain; bone metabolism; osteolytic lesions; DEXA-scans; X-ray radiography
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Zoledronic Acid; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib/Dexamethasone/Zoledronic Acid (Experimental): For this study, Velcade will be administered at the standard dose of 1.3 mg/m2, iv, bolus, on days 1, 4, 8 and 11 of a 21-day cycle.
  Dexamethasone will be administered at a dose of 12 mg/m2 p.o., on days 1-2, 4-5, 8-9 and 11-12 of the same cycle.
  Zoledronic acid will be administered at a dose of 4 mg, iv (15-minute infusion), every 28 days for up to 8 cycles, and then every 28 days for the next 18 months
  Interventions: Drug: Bortezomib; Drug: Zoledronic Acid; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m2, iv, bolus, on days 1, 4, 8 and 11 of a 21-day cycle for up to 8 chemotherapy cycles
  Other Names: Velcade
Drug: Zoledronic Acid — 4 mg, iv, at a 15 min infusion, Day 1 of every cycle for up to 8 cycles, and then every 28 days for the next 18 months
  Other Names: Zometa
Drug: Dexamethasone — 12 mg/m2 p.o. on days 1-2, 4-5, 8-9 and 11-12 of a 21-day cycle for up to 8 chemotherapy cycles

SUMMARY:
The aim of this study is to evaluate the effect of bortezomib in combination with dexamethasone and zoledronic acid on bone mineral density (BMD) and skeletal related events (SREs) in Patients with Multiple Myeloma who Have Relapsed after 1-3 Prior Lines of Therapy

DETAILED DESCRIPTION:
Multiple Myeloma represents a malignant proliferation of plasma cells derived from a single clone. The most common symptom in myeloma, affecting more than 70% of patients at diagnosis, is bone pain. The pain usually involves the back and ribs, and is precipitated by movement. Bone fractures are commonly seen in myeloma patients and may present with persistent localized pain.

VELCADE (bortezomib) is a proteasome inhibitor used for the treatment of multiple myeloma.

VELCADE seems to be the first agent to combine significant anti-myeloma activity and beneficial effects on bone remodeling. Thus, it appears to be a very promising tool for the treatment of myeloma patients.

In this study, a regimen consisting of bortezomib/dexamethasone/zoledronic acid will be used. The rationale for using this regimen is that:

* VELCADE (bortezomib) is indicated for the treatment of relapsed myeloma patients participating in the study and it has also a beneficial effect on biochemical markers of bone formation.
* In phase II studies, the addition of dexamethasone in patients with a suboptimal response to bortezomib alone improved efficacy in relapsed or refractory multiple myeloma patients, without increasing adverse events. Therefore, in this study, the addition of dexamethasone aims at providing the optimal therapy for participating myeloma patients.
* Zoledronic acid, the most potent i.v. bisphosphonate, is used because of its established effect on reducing skeletal related events in patients with multiple myeloma due to its inhibitory effect on osteoclastic bone resorption.

Dosages and timing of dosages are based on current recommendations and guidelines for the treatment of myeloma patients who Have Relapsed after 1-3 Prior Lines of Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple Myeloma who Have Relapsed after 1-3 Prior Lines of Therapy
* Women > 50 years old
* Κarnofsky performance status ≥ 60 (patients with lower performance status due to myeloma bone disease can also be included)
* Measurable disease
* Platelet count >50x10(9)/L
* Neutrophil count >0.75x10(9)/L
* Hemoglobin ≥7.0 g/dL (the use of recombinant human erythropoietin or red blood Hell transfusions to maintain hemoglobin levels above 7.0 g/dL is not an exclusion criterion)
* Serum ALT and AST ≤ 3-fold of upper normal limit
* Serum bilirubin ≤ 2-fold of upper normal limit
* Serum Calcium ≤ 10.5 mg/dL
* Expected survival ≥ 2 months
* Signed informed consent

Exclusion Criteria:

* Presence of another cancer
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Grade 2-4 peripheral neuropathy or neuropathic pain Grade 2 or higher as defined by NCI CTCAE version 3
* Pregnant women > 50 years old or breast-feeding
* Woman > 50 years old capable of becoming pregnant [anyone who has not undergone a hysterectomy, has not had both ovaries removed or has not been post-menopausal for more than 24 months in a row not using adequate contraception
* Known or suspected hypersensitivity or intolerance to bortezomib, boron, mannitol, zoledronic acid, dexamethasone, or heparin (if an indwelling catheter is used)
* Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months prior to first dose of study drug)
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 4, NYHA Classification of Cardiac Disease), uncontrolled angina, pericardial disease, or cardiac amyloidosis
* Acute diffuse infiltrative pulmonary disease
* History of hypotension or patient has decreased blood pressure (sitting systolic blood pressure [SBP] 100 mmHg and/or sitting diastolic blood pressure [DBP] 60 mmHg)
* Patient has received extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks prior to enrolment
* Patient has received any drugs or agents that inhibit (e.g., cimetidine, erythromycin, fluoxetine, ketoconazole, paroxetine) or induce (e.g., carbamazepine, glucocorticoids, phenobarbital, rifampin) CYP2C19 or CYP3A4 within 14 days before the first dose of VELCADE (proton pump inhibitors are allowed)
* Need for therapy with concomitant CYP 3A4 inhibitors (e.g., itraconazole, fluconazole, clarithromycin, erythromycin, norfloxacin, fluvoxamine, cimetidine, indinavir, ritonavir) or inducers (e.g., efavirenz, barbiturates, phenytoin, rifampin, glitazones). Proton pump inhibitors are allowed.
* Patient has received an experimental drug or has used an experimental medical device within 4 weeks prior to the planned start of treatment. Concurrent participation in non-treatment studies is allowed, provided it will not interfere with participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meletios- Athanasios Dimopoulos, Professor, Study Chair — Therapeutic Clinic Department, Faculty of Medicine. University of Athens
Locations (3):
- Greece (3):
  - Department of Clinical Therapeutics, University of Athens School of Medicine, "Alexandra" General Hospital, Athens
  - Department of Hematology & Medical Research, 251 General Air Force Hospital, Athens
  - Department of Hematology, "Theagenion" Cancer Center, Thessaloniki

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib/Dexamethasone/Zoledronic Acid: For this study, Velcade will be administered at the standard dose of 1.3 mg/m2, iv, bolus, on days 1, 4, 8 and 11 of a 21-day cycle.
  Dexamethasone will be administered at a dose of 12 mg/m2 p.o., on days 1-2, 4-5, 8-9 and 11-12 of the same cycle.
  Zoledronic acid will be administered at a dose of 4 mg, iv (15-minute infusion), every 28 days for up to 8 cycles, and then every 28 days for the next 18 months
  Bortezomib: 1.3 mg/m2, iv, bolus, on days 1, 4, 8 and 11 of a 21-day cycle for up to 8 chemotherapy cycles
  Zoledronic Acid: 4 mg, iv, at a 15 min infusion, Day 1 of every cycle for up to 8 cycles, and then every 28 days for the next 18 months
  Dexamethasone: 12 mg/m2 p.o. on days 1-2, 4-5, 8-9 and 11-12 of a 21-day cycle for up to 8 chemotherapy cycles
Period: Overall Study
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Region of Enrollment [Number; unit: participants]
  Greece | 17
BMD [Median (Full Range); unit: T-score] — Bone Mineral Density of the lumbar spine (L1-L4, anteroposterior view) and femoral neck (FN) was measured by Dual Energy X-Absorptiometry scan (DEXA-scan) using a Hologic QDR-1000 scanner
  T-score
    Lumbar spine (L1-L4) | -0.29 [-3.8 to 2.88]
    Femoral neck (FN) | -2.83 [-3.91 to 0.55]
Bone remodelling [Median (Full Range); unit: ng/ml] — Bone remodelling was studied by the measurement of the following serum bone metabolism parameters indices using an enzyme-linked immunosorbent assay (ELISA): i) bone resorption marker C-terminal cross-linking telopeptide of collagen type I (CTX) and ii) bone formation marker [osteocalcin (OC)].
  ng/ml
    CTX | 0.6 [0.3 to 2.1]
    OC | 5.1 [0.1 to 14]
Skeletal survey for osteolytic lesions/fractures [Number; unit: participants] — Skeletal survey was measured using conventional radiography [imaging of the whole skeleton (skull, cervical spine, thoracic spine, lumbar spine, pelvis, humeri, femoral bones)].
  participants | 17
Bone pain [Median (Full Range); unit: units on a scale] — Bone pain was measured with the use of the Visual Analogue Scale. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
  The VAS for Bone Pain was constructed as follows:
  None Mild Moderate Severe Worst possible 1,2 3,4 5,6 7,8 9,10 Lower values are considered to be of a better outcome, higher values are considered to be of a worst outcome.
  units on a scale | 5 [3 to 10]
Bone remodelling [Median (Full Range); unit: U/L] — Bone remodelling was studied by the measurement of the following serum bone metabolism parameters indices using an enzyme-linked immunosorbent assay (ELISA) bone formation marker [bone-specific alkaline phosphatase (bALP)].
  U/L | 15.8 [4.5 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD)
Description: BMD of the lumbar spine (L1-L4, anteroposterior view) and femoral neck (FN) was measured by dual energy X-ray absorptiometry (DXA) using a Hologic QDR-1000 scanner on day 21 of cycle 4 (day 84)
Time Frame: day 84
Population: Out of the 17 patients enrolled 12 patients completed the 8 VD cycles, 2 patients 6 VD cycles (due to peripheral neuropathy), 1 patient 5 VD cycles (and then progressed) and 2 patients died after receiving 1 and 2 VD cycles (respectively)
Measure: Median (Full Range); unit: T-scores
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 15
T-scores
  Lumbar spine (L1-L4) | 0.14 (0.022) [-3.8 to 3.43]
  Femoral neck (FN) | -2.68 (0.009) [-3.6 to 1.5]

2. Secondary Outcome: Bone Mineral Density (BMD)
Description: BMD of the lumbar spine (L1-L4, anteroposterior view) and femoral neck (FN) was measured by Dual Energy X-Absorptiometry scan (DEXA-scan) using a Hologic QDR-1000 scanner on day 21 of cycle 8 (day 168)
Time Frame: day 168
Population: as for outcome 1
Measure: Median (Full Range); unit: T-score
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 15
T-score
  Lumbar spine (L1-L4) | 1.63 (0.01) [-3.37 to 3.5]
  Femoral neck (FN) | -1.44 (0.01) [-3.47 to 1.3]

3. Secondary Outcome: Bone Remodelling
Description: Bone remodelling was studied by the measurement of the following serum indices on day 21 of cycle 4 (day 84) using an enzyme-linked immunosorbent assay (ELISA): i) bone resorption marker C-terminal cross-linking telopeptide of collagen type I (CTX) and ii) bone formation markers [osteocalcin (OC)].
Time Frame: day 84
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 15
ng/ml
  CTX | 0.25 (0.01) [0.04 to 0.9]
  OC | 7.4 [4.2 to 23.8]

4. Secondary Outcome: Bone Remodelling
Description: Bone remodelling was studied by the measurement of the following serum indices on day 21 of cycle 8 (day 168) using an enzyme-linked immunosorbent assay (ELISA): i) bone resorption marker C-terminal cross-linking telopeptide of collagen type I (CTX) and ii) bone formation marker [osteocalcin (OC)].
Time Frame: day 168
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
ng/ml
  CTX | 0.17 (0.01) [0.1 to 0.4]
  OC | 10.2 [1.9 to 40.1]

5. Secondary Outcome: Bone Pain
Description: Bone pain was measured with the use of the Visual Analogue Scale on day 21 of cycle 4 (day 84).
  Bone pain was measured with the use of the Visual Analogue Scale. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
  The VAS for Bone Pain was constructed as follows:
  None Mild Moderate Severe Worst possible 1,2 3,4 5,6 7,8 9,10 Lower values are considered to be of a better outcome, higher values are considered to be of a worst outcome.
Time Frame: On the day 84
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 15
units on a scale | 1.5 (0.01) [1 to 5]

6. Secondary Outcome: Bone Pain
Description: Bone pain was measured with the use of the Visual Analogue Scale on day 21 of cycle 8 (day 168).
  Bone pain was measured with the use of the Visual Analogue Scale. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
  The VAS for Bone Pain was constructed as follows:
  None Mild Moderate Severe Worst possible 1,2 3,4 5,6 7,8 9,10 Lower values are considered to be of a better outcome, higher values are considered to be of a worst outcome.
Time Frame: On the day 168
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
units on a scale | 0.3 (0.01) [0 to 3]

7. Secondary Outcome: Skeletal Survey for New Osteolytic Lesions/Fractures
Description: Skeletal survey was measured using conventional radiography [imaging of the whole skeleton (skull, cervical spine, thoracic spine, lumbar spine, pelvis, humeri, femoral bones)] on day 21 of cycle 8 (day 168)
Time Frame: day 168
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
participants | 0

8. Secondary Outcome: Skeletal Survey for New Osteolytic Lesions/Fractures
Description: Skeletal survey was measured using conventional radiography [imaging of the whole skeleton (skull, cervical spine, thoracic spine, lumbar spine, pelvis, humeri, femoral bones)] every 6 months for up to 18 months
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
participants | 0

9. Secondary Outcome: New Skeletal-related Events (SRE: Pathologic Fractures, Need for Bone Radiation Therapy or Surgery)
Description: New Skeletal-related events (SRE: pathologic fractures, need for bone radiation therapy or surgery) following 8 cycles (day 168) of therapy
Time Frame: day 168
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
participants | 0

10. Secondary Outcome: New Skeletal-related Events (SRE: Pathologic Fractures, Need for Bone Radiation Therapy or Surgery)
Description: New Skeletal-related Events (SRE: Pathologic Fractures, Need for Bone Radiation Therapy or Surgery) after 18 months post VD
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
participants | 0

11. Secondary Outcome: Bone Remodelling
Description: Bone remodelling was studied by the measurement of the following serum indices on day 21 of cycle 4 (day 84) using an enzyme-linked immunosorbent assay (ELISA) bone formation marker [bone-specific alkaline phosphatase (bALP)].
Time Frame: day 84
Population: as for outcome 1
Measure: Median (Full Range); unit: U/L
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 15
U/L | 22.5 [9.9 to 35]

12. Secondary Outcome: Bone Remodelling
Description: Bone remodelling was studied by the measurement of the following serum indices on day 21 of cycle 4 (day 84) using an enzyme-linked immunosorbent assay (ELISA): bone formation marker [bone-specific alkaline phosphatase (bALP) ].
Time Frame: day 168
Population: as for outcome 1
Measure: Median (Full Range); unit: U/L
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Number analyzed (Participants) | 12
U/L | 24.8 [14 to 35]

ADVERSE EVENTS:
Arm/Group | Bortezomib/Dexamethasone/Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib/Dexamethasone/Zoledronic Acid (N=17)
Death due to cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Death due to thrombocytopenia grade IV (Blood and lymphatic system disorders) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 1 (1)
infection of lower respiratory (Infections and infestations) | 2 (2)
bacteraemia (Infections and infestations) | 1 (1)
anemia and thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No